CLINICAL TRIAL: NCT02807012
Title: Nursing Home Care Educational Intervention for Family Caregivers of Older Adults Post Stroke
Brief Title: Nursing Home Care Intervention Post Stroke
Acronym: SHARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16-0181
Record Dates: First submitted 2016-06-03; First posted 2016-06-21 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-03

CONDITIONS: Stroke
Keywords: Home care services; Nursing; Clinical trial; Geriatric nursing; Family caregiver; Aged
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nursing educational intervention (Experimental): The intervention will consist in three home visits (14, 21, 30 days after discharge) by nurses to family caregivers. The nurses will give verbal information and printed materials related to the care of older adults por stroke.
  Interventions: Other: Nursing educational intervention
- Usual care (No Intervention): The family caregivers won't receive the home visits and could have or not the usual care guidelines provide by health services that have access.

INTERVENTIONS:
Other: Nursing educational intervention — The nursing educational intervention by home visits will consist in three home visits by nurses until 14, 21 and 30 days after discharge to the intervention group. The nurses will give verbal information to family caregiver related to the care of elderly with stroke based on protocol with orientation related: information about stroke; emotional support; how to access health services; nutrition; airway; hygiene; positioning and transferring; prevent falls; dress/undress; medications; physiological eliminations; skin care. Furthermore, nurses will give some printed materials that contain orientations related to the care.
  The control group could have ou not the usual care guidelines provide by health services that have access.
  Arms: Nursing educational intervention

SUMMARY:
Associated with the worsening of functional capacity of older adult and the lack of guidance on how to care of them after stroke, the family caregiver starts to fell burden related to the care, and the quality of life was affected by that burden. Besides that, the older adult began to use more frequently health services and had more hospitalizations by preventable conditionals with adequate care.

The aim of this study is to evaluate the effectiveness of educational interventions of care at home provide by nurses to family caregivers of older adult with stroke after hospital discharge, compared with usual care guidelines or no guidance, in one month follow up. The family caregivers of older adults post stroke with the first functional sequel from the Clinical Hospital of Porto Alegre (HCPA) will participate in the study.

The intervention will involve the systematic monitoring of nurses through home visits (HVs) during one month. Thus, will instrumentalize the family caregiver to care of older adult with stoke according the protocol developed in a research group and the needs of care of them. The control group won't receive the home visits and could have or not the usual care guidelines provide by health services that have access.

DETAILED DESCRIPTION:
Associated with the worsening of functional capacity of older adult and the lack of guidance on how to care of them after stroke, the family caregiver starts to fell burden related to the care and the quality of life was affected by that burden. Besides that, the older adult began to use more frequently health services and had more hospitalizations by preventable conditionals with adequate care.

The aim of this study is to evaluate the effectiveness of educational interventions of care at home provide by nurses to family caregivers of older adult with stroke after hospital discharge, compared with usual care guidelines or no guidance, in one month follow up. The family caregivers of older adults post stroke with the first functional sequel from the Clinical Hospital of Porto Alegre (HCPA) will participate in the study. The randomization will be through the randomization list created by web page randomization.com.

The intervention will involve systematic monitoring of nurses through home visits (HVs) during one month. Thus, will instrumentalize the family caregiver to care of older adult with stoke according the protocol developed in a research group and the needs of care of them. The control group won't receive the HVs and could have or not the usual care guidelines provide by health services that have access.

Will be collect the identification, social and demographics data of the older adults and the caregivers at the moment of hospital discharge. Therefore, will be collect the clinical data of the older adults. After discharge and at the older adult's home, will be realized the first home visit (1ª HV) to all older adults and caregivers included in the study and will be applied to the family caregiver the Caregiver Burden Scale and the instrument WHOQOL-BREF that analyse the quality of life. Also, will be applied the Measure of Functional Independence (MIF) to identify the independence level of the older adults and the needs of care. In this moment, will be randomized by an extern member of research group through telephone contact. After this first HV, the older adults and caregivers included in the intervention group will received more three HVs, until 14, 21 and 30 days after discharge, respectively, by a pair of interventional nurses.

The control group won't receive the home visits by nurses, but could have or not the usual care guidelines provide by health services that have access.

All older adults and caregivers included in the study will received a fifth HV until 60 days after discharge. In this last HV will be applied to family caregiver the Caregiver Burden Scale and the instrument WHOQOL-BREF. In addition, will be applied a questionnaire related older adult's utilization of health services and rehospitalizations during this time and the MIF.

ELIGIBILITY:
Inclusion Criteria:

* Family caregivers of older adults from the Special Care Unit - stroke (SCU-Stroke) at the moment of discharge;
* Older adults with diagnosis of stroke with the first sequel identified by minimum score of 2 points from the ranking scale;
* Older adults who live until 20 kilometers from HCPA;
* Caregiver will be a family member with consanguineous relationship or not;
* Caregiver will be responsible for the most part of the older adult's care;
* Caregiver without payment;
* Caregiver with 18 year old or more.

Exclusion Criteria:

* Older adults who live in a Long Term Care Services;
* Older adults who will be included in a governmental program for Home Care Service;
* Caregivers who don't accept receive the HV by nurses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
The family caregiver's burden of care analyzed by Caregiver Burden Scale | 2 months
  The family caregiver burden of care will be analyzed by Caregiver Burden Scale.

SECONDARY OUTCOMES:
The family caregiver's quality of life analyzed by instrument WHOQOL-BREF | 2 months
  The family caregiver quality of life will be analyzed by instrument WHOQOL-BREF.
The elderly's functional capacity | 2 months
  The elderly functional capacity will be analyzed by the instrument Measure of Functional Independence
The elderly's health service utilization | 2 months
  The elderly health service utilization will be assessed by an questionnaire developed for this study. The answers will be yes or not and analyzed quantitatively.
The elderly's rehospitalization | 2 months
  The elderly rehospitalization will be assessed by an questionnaire developed for this study. The answers will be yes or not and analyzed quantitatively.
The quality of life of family caregiver with 60 years old or older analyzed by instrument WHOQOL-OLD | 2 months
  The family caregiver quality of life will be analyzed by instrument WHOQOL-OLD

CONTACTS AND LOCATIONS:
Overall Officials: Lisiane MG Paskulin, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bierhals CCBK, Dal Pizzol FLF, Low G, Day CB, Santos NOD, Paskulin LMG. Quality of life in caregivers of aged stroke survivors in southern Brazil: Arandomized clinical trial. Rev Lat Am Enfermagem. 2023 Jan-Dec;31:e3657. doi: 10.1590/1518-8345.5935.3657. PMID 36722630
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Day CB, Bierhals CCBK, Mocellin D, Predebon ML, Santos NO, Dal Pizzol FLF, Fuhrmann AC, Aires M, Paskulin LMG. Nursing Home Care Intervention Post Stroke (SHARE) 1 year effect on the burden of family caregivers for older adults in Brazil: A randomized controlled trial. Health Soc Care Community. 2021 Jan;29(1):56-65. doi: 10.1111/hsc.13068. Epub 2020 Jun 30. PMID 32602588
- [Derived] Bierhals CCBK, Day CB, Mocellin D, Santos NOD, Predebon ML, Pizzol FLFD, Fuhrmann AC, Medeiros GG, Aires M, Paskulin LMG. Use of health services by elderly people post-stroke: a randomized controlled trial. Rev Gaucha Enferm. 2019 Dec 2;41(spe):e20190138. doi: 10.1590/1983-1447.2020.20190138. eCollection 2020. English, Portuguese. PMID 31800798
- [Derived] Day CB, Bierhals CCBK, Santos NOD, Mocellin D, Predebon ML, Dal Pizzol FLF, Paskulin LMG. Nursing home care educational intervention for family caregivers of older adults post stroke (SHARE): study protocol for a randomised trial. Trials. 2018 Feb 9;19(1):96. doi: 10.1186/s13063-018-2454-5. PMID 29426361